CLINICAL TRIAL: NCT01966939
Title: Influences of Types of Skull Surgery on Temporomandibular Joint Performance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201106049RC; UN101-005 (Other Grant/Funding Number: NTUH)
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Craniotomy; Craniectomy
Keywords: craniotomy; craniectomy; temporalis; TMJ; mastication; QoL

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgery: Craniotomy or Craniectomy
- Control: age, gender and teeth condition matched

SUMMARY:
There are two purposes on this study:

- to investigate the effect of craniectomy and craniotomy on temporomandibular joint TMJ) movement, function and quality of life (QoL)

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* post-craniotomy or post-craniectomy
* able to follow order

Exclusion Criteria:

* severe orofacial injury
* severe teeth loss
* significant changes of occlusion

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects received craniotomy or craniectomy and age, gender and teeth condtion matched control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Jaw movement | within 1 year after surgery
Jaw Functional Limitation Scale | within 1 year after surgery
Bite force | within 1 year after surgery
WHOQOL-BREF Taiwanese Version | within 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan